CLINICAL TRIAL: NCT02035384
Title: A Multi-centre Non-interventional Study of Safety and Efficacy of Turoctocog Alfa (rFVIII) During Long-Term Treatment of Severe and Moderately Severe Haemophilia A (FVIII =<2%)
Brief Title: Safety and Efficacy of Turoctocog Alfa During Long-Term Treatment of Severe and Moderately Severe Haemophilia A
Acronym: guardian™ 5
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7008-3553; U1111-1126-0353 (Other: WHO); ENCEPP/SDPP/5501 (Registry Identifier: EU PAS)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients
  Interventions: Drug: turoctocog alfa

INTERVENTIONS:
Drug: turoctocog alfa — Patients will be treated with commercially available turoctocog alfa as prescribed by the treating physician in clinical daily practice and preferably according to the label for turoctocog alfa in the respective countries.

SUMMARY:
This study is conducted in Europe, and North and South America. The aim of this study is to provide additional documentation of the immunogenicity, and obtain additional clinical data, of turoctocog alfa in the setting of normal clinical practise in patients previously treated with a factor VIII agent (FVIII).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedure related to recording of data according to the protocol
* Previously FVIII treated (150 exposure days at the time of first dosing with turoctocog alfa) male patients with the diagnosis of severe and moderately severe haemophilia A (FVIII below or equal to 2%)
* The decision to initiate treatment with commercially available turoctocog alfa has been made by the patient/parent and the patient's treating physician before and independently from the decision to include the patient in this study
* A negative FVIII inhibitor test obtained not more than four weeks prior to first dosing with turoctocog alfa

Exclusion Criteria:

* Contraindications for use according to the approved product information text (US Package insert (PI), European Summary of Product Characteristics (SmPC), or corresponding local prescribing information)
* Treatment with any investigational drug within 30 days prior to enrolment into the study
* Previous participation in any clinical trial with turoctocog alfa
* Treatment with other FVIII products after initiation of treatment with turoctocog alfa

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Previously FVIII treated (more than 150 exposure days) patients with severe and moderately severe haemophilia A with FVIII below or equal to 2%.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Incidence rate of FVIII inhibitors (at least 0.6 Bethesda Units (BU) for central laboratory analyses, or above the specific local laboratory reference range) represented as the percentage of patients developing inhibitors | Within approximately 7 years

SECONDARY OUTCOMES:
Number of adverse reactions reported | During approximately 7 years
Number of serious adverse reactions reported | During approximately 7 years
Haemostatic effect of turoctocog alfa in the treatment of bleeds as assessed by the patient or the physician according to a predefined four point scale: Excellent, Good, Moderate, or None | Within approximately 7 years
Haemostatic effect of turoctocog alfa during surgical procedures as assessed by an evaluation according to a predefined four point scale: Excellent, Good, Moderate, or None | Within approximately 7 years
Annualised bleeding rate for patients using turoctocog alfa for preventive treatment | Within approximately 7 years
Annualised bleeding rate for patients using turoctocog alfa for on-demand treatment | Within approximately 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (41):
- United States (6):
  - Novo Nordisk Investigational Site, Mobile, Alabama
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
- Austria (2):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Linz
- Novo Nordisk Investigational Site, Brno, Czechia
- France (5):
  - Novo Nordisk Investigational Site, Bordeaux
  - Novo Nordisk Investigational Site, Montmorency
  - Novo Nordisk Investigational Site, Rennes
  - Novo Nordisk Investigational Site, Saint-Etienne
  - Novo Nordisk Investigational Site, Strasbourg
- Germany (8):
  - Novo Nordisk Investigational Site, Braunschweig
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Frankfurt am Main
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Leipzig
  - Novo Nordisk Investigational Site, Mörfelden-Walldorf
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Münster
- Novo Nordisk Investigational Site, Athens, Greece
- Hungary (3):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Mohács
- Italy (5):
  - Novo Nordisk Investigational Site, Castelfranco Veneto
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Palermo
- Netherlands (2):
  - Novo Nordisk Investigational Site, The Hague
  - Novo Nordisk Investigational Site, Utrecht
- Novo Nordisk Investigational Site, Warsaw, Poland
- Slovakia (2):
  - Novo Nordisk Investigational Site, Banská Bystrica
  - Novo Nordisk Investigational Site, Košice
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- Novo Nordisk Investigational Site, Barcelona, Spain
- Sweden (2):
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
- Novo Nordisk Investigational Site, Zurich, Switzerland

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com